CLINICAL TRIAL: NCT05364450
Title: Acceptance and Commitment Therapy for Fear of Recurrence in Breast Cancer Survivors
Brief Title: Facilitating Adaptive Coping With Fear of Recurrence Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other); Eskenazi Health (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shelley Johns, Associate Professor of Medicine, Research Scientist, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 11066; R01CA255480 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasm; Breast Cancer; Breast Carcinoma; Malignant Neoplasm of Breast; Cancer of Breast; Mammary Neoplasms, Human; Human Mammary Carcinoma; Malignant Tumor of Breast; Mammary Cancer; Mammary Carcinoma, Human; Anxiety; Fear
Keywords: Fear of Cancer Recurrence; Fear of Cancer Return; Breast Cancer Survivor; Breast Cancer Remission
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: An external statistician will create the randomization sequence. An unblinded research manager will maintain the randomization sequence and randomization assignment for each participant in password-protected databases not accessible by the study team. All study personnel, including the study's principal investigator (PI), biostatistician, data manager, research coordinator (RC), and research assistants (RAs), will be blind to the randomization sequence. The PI, research manager, interventionists, and intervention supervisors will be the only individuals privy to participants' randomization assignments. The study RC, RAs (including outcome assessors), and the study biostatistician and data manager will remain blind to participants' random assignments for the trial's duration to enhance rigor and reduce the risk of outcome expectancy and other biases. Participants will be blind to study hypotheses, yet will be aware of their assignment to a 6-session versus single-session intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (EUC) (Active Comparator): The EUC group will meet for a single 90-minute coaching session via Zoom Health.
  Interventions: Behavioral: Enhanced Usual Care
- Acceptance Commitment Therapy (ACT) (Active Comparator): The ACT group will meet for 90-minute sessions via Zoom Health weekly for 6 weeks.
  Interventions: Behavioral: Acceptance Commitment Therapy
- Cognitive Behavioral Therapy (CBT) (Active Comparator): The CBT group will meet for 90-minute sessions via Zoom Health weekly for 6 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Enhanced Usual Care — Interventionists will provide a brief explanation of the intervention and coaching to the group on how to utilize the resources provided. Prior to the single session group, EUC participants will have received a workbook with the National Cancer Institute's "Facing Forward: Life After Cancer Treatment" booklet on maximizing quality of life during cancer survivorship and the American Society of Clinical Oncology's "Guide to Cancer Survivorship."
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)
Behavioral: Acceptance Commitment Therapy — Interventionists will support participants in adopting a psychologically flexible posture toward FCR through six interdependent processes of change - acceptance, cognitive defusion, mindfulness, perspective taking, values, and committed action. During ACT sessions, participants will learn to respond adaptively to FCR by being more fully aware of thoughts, feelings, and bodily sensations without judging or attempting to control or avoid them. Participants will also clarify their deeply-held values and set action goals in alignment with their values.
  Other Names: ACT
  Arms: Acceptance Commitment Therapy (ACT)
Behavioral: Cognitive Behavioral Therapy — Interventionists will provide psycho-education on the cognitive behavioral model of FCR and assist participants in changing unhelpful thinking patterns and maladaptive behaviors linked to FCR. Session topics will include FCR triggers, behavioral experiments to reduce FCR-perpetuating safety behaviors, and pleasant events scheduling. Interventionists will also provide evidence-based information on behaviors that may reduce recurrence risk (e.g., achieving a healthy weight, physical activity, cancer surveillance).
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
Fear of cancer recurrence (FCR) is a highly prevalent, disruptive, and under-treated problem for breast cancer survivors. This randomized controlled trial will test the efficacy of group-based Acceptance and Commitment Therapy compared to Cognitive Behavioral Therapy and enhanced usual care for breast cancer survivors suffering from FCR while examining its cost-effectiveness and the mechanisms by which the intervention may work. Study findings will guide the future care of breast cancer survivors with FCR.

DETAILED DESCRIPTION:
The primary objective of this 3-arm randomized control trial (RCT) is to build on the investigators' pilot work by testing the impact of Acceptance Commitment Therapy (ACT) on FCR. The investigators will randomly assign up to 375 early-stage Breast Cancer Survivors (BCS; for at least 300 study completers after attrition) who have finished primary cancer treatment and who report clinically significant FCR to: (1) group-based ACT (6 weekly 1.5-hour videoconference sessions), (2) group-based Cognitive Behavioral Therapy (CBT; 6 weekly 1.5-hour videoconference sessions), or (3) Enhanced Usual Care (EUC; a single 90-minute videoconference coaching session with self-administered readings). Outcomes will be assessed at baseline and at 2, 6, and 12 months; additionally, potential theory-driven mediators of the ACT intervention's effects on key outcomes will be analyzed at these time points and at intervention midpoint. Cost-effectiveness of each intervention will be assessed.

Specific Aims are to: (1) test the efficacy of group-based ACT compared to CBT and EUC on FCR (primary outcome) and anxiety, depressive symptoms, post-traumatic stress, avoidant coping, fatigue, sleep disturbance, and quality of life (secondary outcomes) in BCS with clinical FCR; (2) to examine changes in psychological flexibility as a mediator of ACT's effect on FCR; and (3) to perform comparative assessments of ACT, CBT, and EUC to determine the cost-effective intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years old.
* Patient has been diagnosed with stage I-IIIA breast cancer without evidence of distant disease at time of study entry.
* Patient has completed surgery, radiation therapy, chemotherapy, and/or biologic therapy ≤5 years prior (ongoing endocrine therapy is allowed).
* Patient has clinically significant FCR (FCR-7 score ≥17 at screening).
* Patient is willing to be randomized into any of the 3 arms of the trial and attend a 6-week videoconference group if randomly assigned to ACT or CBT and a single videoconference group if randomly assigned to EUC.
* Patient is able to speak and read English

Exclusion Criteria:

* Patient has a previous cancer diagnosis besides breast (non-melanoma skin cancer or melanoma in situ is allowed).
* Patient is currently participating in ACT, CBT, formal mindfulness meditation training, the "Mobile Device CBT for Chemotherapy-Related Cognitive Dysfunction: A Multi-Center Randomized Controlled Trial," the "Thinking and Living With Cancer" study, or any other research study that has the potential to skew results of this study or the study in which the person is participating.
* Patient has co-morbidities, medications, or deficits that would impair participation in any of the 3 groups (ACT, CBT or EUC), including: history of stroke, encephalitis, traumatic brain injury/surgery, Alzheimer's disease, or other dementia; severe depressive symptoms (PHQ-2 score ≥5 at screening); active substance abuse or uncontrolled bipolar disorder, psychosis, or schizophrenia; obvious hearing and/or communicative disability.
* Patient has opted out of pre-screening for research studies (sometimes noted in the electronic medical record)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Fear of Cancer Recurrence from Baseline | given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 43-item Fear of Cancer Recurrence Inventory (FCRI) includes triggers, psychological distress, coping strategies, reassurance seeking, insight, severity, and functional impairments subscales. Each item is rated on a scale from 0 (never, not at all, or I don't think about it) to 4 (all the time or a great deal), participants indicate the extent to which they are fearful, with higher scores indicating greater FCR.

SECONDARY OUTCOMES:
Change in Fear of Cancer Recurrence Questionnaire - 7 (FCR-7) from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 7-item FCR-7 assesses anxiety, worry, and strong feelings associated with cancer recurrence, coupled with items assessing cognitive and behavioral responses to FCR. The first six items are on a scale from 1 (not at all) to 5 (all the time). The seventh item assesses the extent to which worry about getting cancer again intrudes on thoughts and activities on a 0 (not at all) to 10 (great deal) scale. Higher scores indicate greater FCR.
Change in Concerns about Recurrence (CARS) from Baseline | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 4-item Concerns About Recurrence Scale includes frequency, potential for upset, consistency, and intensity of fears on a 1-4 scale. Higher scores indicate greater FCR.
Fear of Cancer Recurrence Global Anchor | Given at 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  Participants will be asked "Overall, since starting your assigned study program, is your fear of cancer recurrence worse, about the same, or better?" Those rating their fear of cancer recurrence as "better" are then asked if their fear is "a little better," "somewhat better," "moderately better," "a lot better," or "completely better".
Change in Anxiety Symptoms from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 7-item Generalized Anxiety Disorder Scale (GAD-7) assesses how often in the past two weeks participants have been bothered by symptoms of anxiety on a 0 (not at all) to 3 (nearly everyday) scale, with higher scores indicating greater anxiety.
Change in Anxiety from Baseline | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety measure assesses how often participants felt various symptoms of anxiety in the past 7 days on a 1 (never) to 5 (always) scale, with higher scores indicating greater anxiety.
Change in Post-Traumatic Stress Symptoms from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 22-item Impact of Events Scale-Revised (IES-R) assesses post-traumatic distress on a 0 (not at all) to 4 (extremely) scale, with higher scores indicating greater post traumatic distress.
Change in Depressive Symptoms from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 8-item Patient Health Questionnaire (PHQ-8) depression scale assesses how often participants have been bothered with symptoms of depression over the past two weeks on a 0 (not at all) to 3 (nearly everyday) scale, with higher scores indicating greater depressive symptomatology.
Change in Depression from Baseline | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 4-item PROMIS Depression measure assesses how often participants felt various symptoms of depression in the past 7 days on a 1 (never) to 5 (always) scale, with higher scores indicating greater depression severity.
Change in Fatigue from Baseline | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 4-item PROMIS Fatigue measure assesses how often participants felt various symptoms of fatigue in the past 7 days on a 1 (not at all) to 5 (very much) scale, with higher scores indicating greater fatigue severity.
Change in Sleep Disturbance from Baseline | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 4-item PROMIS Sleep Disturbance measure assesses how often participants experienced aspects of sleep disturbance in the past 7 days on a 1 (not at all) to 5 (very much) scale, with higher scores indicating greater sleep disturbance.
Change in Coping from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 28-item Brief COPE assesses how often participants have been utilizing a series of coping strategies since their cancer diagnosis on a 1 (I haven't been doing this at all) to 4 (I have been doing this a lot) scale, with higher scores indicating greater use of the coping strategy.
Change in Quality of Life from Baseline | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 10-item PROMIS Global Health measure assesses mental and physical health. The first nine items are on a 1 (poor or not at all) to 5 (excellent or completely) scale. The tenth item assesses average pain on a 0 (no pain) to 10 (worst pain imaginable) scale and is reverse scored. Higher scores are indicative of better global health.

OTHER OUTCOMES:
Change in Health-Related Quality of Life | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  EuroQoL Five Dimensions Questionnaire (EQ-5D-5L) is a standardized non-disease specific instrument used to estimate 'utilities' for cost-effectiveness analyses. Consists of 5 items assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 1-5 scale. An additional item asks respondents to assess overall health on a 0 (worst health imaginable) to 100 (best health imaginable) scale. This measure will be used in cost effectiveness analysis.
Direct and indirect medical and non-medical costs | Given at baseline (T1), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  Medical and non-medical costs are measure over the past 4 weeks using the validated Treatment Inventory of Costs in Patients with Psychiatric Disorders (TiC-P). The first part of the TiC-P assesses frequency of use of various types of health care resources. The second part is an adaptation of the Short Form of the Health and Labor Questionnaire. This measure will be used in cost effectiveness analysis.
Change in Psychological Flexibility | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 18-item Cancer Acceptance and Action Questionnaire is a validated measure of cancer-related psychological flexibility, with items rated on a 1 (never true) to 7 (always true) scale. Lower scores indicate greater psychological flexibility. This measure will be used in mediator analysis.
Change in Mindfulness | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 10-item Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) comprehensively assesses mindfulness processes including attention, present-focused awareness, and acceptance/non-judgment. Items are rated on a 1 (rarely or not at all) to 4 (almost always) scale, with higher scores indicating greater mindfulness. This measure will be used in mediator analysis.
Change in Commitment and Behavior Change | Given at baseline (T1), intervention midpoint (T-Mid), 2 months post-baseline (T2), 6 months post-baseline (T3), and 12 months post-baseline (T4)
  The 5-item Value Progress subscale of the Valuing Questionnaire assesses progress in living consistently with personal values. Items are rated on a 0 (not at all true) to 6 (completely true) scale, with higher scores indicating greater values-consistent living. This measure will be used in mediator analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A Johns, PsyD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University-Purdue University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH funded study - public database
Supporting Information: Study Protocol, SAP
Time Frame: A completed data set will be available in approximately May of 2025. De-identified data will be made available to qualified investigators within 6 months of acceptance of the manuscript describing major outcomes.
Access Criteria: Investigators who request to use the de-identified dataset will be required to obtain Institutional Review Board approval and sign a data use agreement before data will be released. The data use agreement must include the following commitments: (1) use of the data will be only for their scholarly research purposes; (2) the data will be secured using appropriate computer technology (e.g., encryption, password protection) and confidentiality of the data will be maintained; (3) the data will be destroyed or returned after analyses are complete; and (4) compliance with Indiana University's Human Subjects Protection Program institutional requirements regarding handling of study data.

DOCUMENTS (1):
  • Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT05364450/ICF_000.pdf